CLINICAL TRIAL: NCT01636401
Title: Efficacy and Safety of 400 μg Twice Daily of Aclidinium Bromide vs. Placebo When Administered to Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_EKL001
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

ARMS (2):
- aclidinium bromide (Active Comparator)
  Interventions: Drug: aclidinium bromide 400 μg
- Placebo (Placebo Comparator)
  Interventions: Drug: aclidinium bromide placebo

INTERVENTIONS:
Drug: aclidinium bromide 400 μg
  Arms: aclidinium bromide
Drug: aclidinium bromide placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to observe the Efficacy and safety of 400 μg twice daily of aclidinium bromide vs. placebo when administered to patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stable moderate to severe COPD as defined by GOLD (the Global Initiative for Chronic Obstructive Lung Disease) guidelines(http://www.goldcopd.org); a postbronchodilator FEV1/forced vital capacity [FVC] ratio < 70% and FEV1 ≥ 30% to <80% of the predicted value.
* Current or former cigarette smokers with a smoking history of at least 10 pack-years.

Exclusion Criteria:

* History or current diagnosis of asthma
* Patients who have been hospitalized for an acute COPD exacerbation within 3 months prior to Visit 1
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the 6 weeks before Visit 1.
* Patients with any clinically significant respiratory conditions other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in morning predose (trough) FEV1 | Week 12

SECONDARY OUTCOMES:
Change from baseline to Week 12 in peak FEV1 | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee SH, Lee J, Yoo KH, Uh ST, Park MJ, Lee SY, Kim JY, Kim DK, Kim SJ, Lee KH, Yoo CG. Efficacy and safety of aclidinium bromide in patients with COPD: A phase 3 randomized clinical trial in a Korean population. Respirology. 2015 Nov;20(8):1222-8. doi: 10.1111/resp.12641. Epub 2015 Sep 15. PMID 26370136